CLINICAL TRIAL: NCT01415154
Title: A 12-Month Prospective Randomized Dual-Arm Pilot Study of Maintenance NeuroStar Transcranial Magnetic Stimulation (TMS) in Patients With Major Depressive Disorder
Brief Title: Maintenance NeuroStar Transcranial Magnetic Stimulation (TMS) in Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44-03001-000
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: TMS; Major Depressive Disorder; NeuroStar TMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Scheduled Treatment Arm (Active Comparator): Following completion of the efficacy assessments at Week 6, One NeuroStar TMS session every four week and TMS reintroduction as needed for clinical deterioration.
  Interventions: Device: NeuroStar TMS
- Monthly Observational Follow up Arm (No Intervention): Following completion of the efficacy assessments at Week 6, Office follow up every 4 week and NeuroStar TMS reintroduction as needed for clinical deterioration.

INTERVENTIONS:
Device: NeuroStar TMS — NeuroStar TMS treatmant - 120% of Observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/sessions for 6 days. 3 treatments in taper week 1, 2 treatments in taper week 2 and 1 treatment in taper week 3.
  Arms: Scheduled Treatment Arm

SUMMARY:
The purpose of this study is to evaluate the efficacy of scheduled maintenance Transcranial Magnetic Stimulation (TMS) treatment compared to on-demand TMS treatment for symptomatic worsening in patients who have shown a clinical response to acute TMS treatment.

DETAILED DESCRIPTION:
This is a 12-month maintenance treatment study for patients who have responded to a 6 week course of acute TMS treatment for major depressive disorder (MDD). The study will seek to assess the change in depressive symptomatology across the duration of maintenance treatment using observer and self-administered efficacy measures. Describe the efficacy of TMS re-introduction in patients not receiving maintenance pharmacotherapy who show a recurrence of depressive symptoms. Assess the safety and durability of acute TMS therapy followed by maintenance TMS treatment for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis by DSM-IV criteria for Major Depressive Episode, single episode or recurrent course of illness, with the additional stipulation of a duration for this episode of ≥ 4 weeks and CGI-S ≥ 4.
* Duration of current episode of depression ≤ 3 years (the definition of an episode is demarcated by a period of ≥ 2 months when the patient did not meet full criteria for the DSM-IV definition of Major Depressive Episode.
* Capable and willing to provide informed consent.
* Signed HIPAA authorization.
* Able to adhere with the treatment schedule, and withdrawal of ongoing pharmacotherapy.
* If currently taking antidepressant pharmacotherapy, must be clinically appropriate to discontinue treatment with those agents.

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption).
* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated):

  * Depression secondary to a general medical condition, or substance- induced;
  * Seasonal pattern of depression as defined by DSM-IV;
  * History of substance abuse or dependence within the past year except nicotine and caffeine);
  * Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes;
  * Bipolar disorder;
  * Eating disorder (current or within the past year);
  * Obsessive compulsive disorder (lifetime); or
  * Post-traumatic stress disorder (current or within the past year).
* An Axis II Personality Disorder, which in the judgment of the Investigator may hinder the patient in completing the procedures required by the study protocol.
* Individuals with a clinically defined neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure;
  * Space occupying brain lesion;
  * History of cerebrovascular accident;
  * Transient ischemic attack within two years;
  * Cerebral aneurysm;
  * Dementia;
  * Parkinson's disease;
  * Huntington's chorea;
  * Multiple sclerosis.
* Increased risk of seizure for any reason, including but not limited to prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for ≥ 5 minutes.
* History of treatment with Vagus Nerve Stimulation.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Brock, MD, Study Director — Neuronetics
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Premier Psychiatric Group, L.L.C., Lincoln, Nebraska
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Center for Anxiety and Depression, Mercer Island, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 patients did not continue to randomization
  A) 12 failed randomization criteria:
  Acute phase endpoint HAMD17 total score <15 and had more than 25% improvement in total score HAMD17 compared with baseline
  B) 2 Patients moved
  C) 2 patients had inadequate response during Acute Phase
  D) 1 patient refused to return
  E) 1 patient had an unrelated panic attack
Groups:
- Monthly Observational Follow up Arm: Following completion of the efficacy assessments at Week 6, Office follow-up visit once every 4 week and TMS reintroduction as needed for clinical deterioration.
Period: Overall Study
Arm/Group | Scheduled Treatment Arm | Monthly Observational Follow up Arm
Started | 23 | 26
Completed | 10 | 6
Not Completed | 13 | 20
Not completed — Lack of Efficacy | 4 | 5
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Lost to Follow-up | 1 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Satisfactory Response | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Scheduled Treatment Arm: 3 Week TMS taper, clinical assessments and one NeuroStar TMS session every 4th week of block and TMS reintroduction as needed for clinical deterioration.
  NeuroStar TMS: NeuroStar TMS treatmant - 120% of Observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/sessions for 6 days. 3 treatments in taper week 1, 2 treatments in taper week 2 and 1 treatment in taper week 3.
- Monthly Observational Follow up Arm: 3 Week TMS Taper, clinical assessments and office follow up every 4th week of block and NeuroStar TMS reintroduction as needed for clinical deterioration.
  NeuroStar TMS: NeuroStar TMS treatmant - 120% of Observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/sessions for 6 days. 3 treatments in taper week 1, 2 treatments in taper week 2 and 1 treatment in taper week 3.
- Total: Total of all reporting groups
Arm/Group | Scheduled Treatment Arm | Monthly Observational Follow up Arm | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.3) | 49.0 (9.8) | 48.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Maintaining a Sustained Response Throughout a 12 Month Maintenance Treatment Phase.
Description: Sustained response is defined as not requiring TMS reintroduction at every observation point during the maintenance phase.
Time Frame: 12 month evaluation
Measure: Count of Participants; unit: Participants
Groups:
- Monthly Observational Follow up Arm: Following completion of the efficacy assessments at Week 6, Office follow-up visit once every 4 week and TMS reintroduction as needed for clinical deterioration.
  NeuroStar TMS: NeuroStar TMS treatmant - 120% of Observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/sessions for 6 days. 3 treatments in taper week 1, 2 treatments in taper week 2 and 1 treatment in taper week 3.
Arm/Group | Scheduled Treatment Arm | Monthly Observational Follow up Arm
Number analyzed (Participants) | 23 | 26
Participants | 5 | 4

2. Secondary Outcome: Average Time to First Reintroduction of TMS Between the Two Maintenance Treatment Arms.
Description: Change in depressive symptomatology will be assessed across the duration of maintenance treatment using observer and self-administered efficacy measures.
Time Frame: 12 Month evaluation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Scheduled Treatment Arm | Monthly Observational Follow up Arm
Number analyzed (Participants) | 23 | 26
days | 103.5 (61.3) | 97.8 (59.1)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Scheduled Treatment Arm | Monthly Observational Follow up Arm
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes